CLINICAL TRIAL: NCT00132756
Title: Liposomal Doxorubicin and Estramustine Phosphate: A Phase II Study in Taxane Resistant, Hormone Refractory Advanced Prostate Cancer
Brief Title: Liposomal Doxorubicin and Estramustine Phosphate: Study in Taxane Resistant, Hormone Refractory Advanced Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Morton Plant Mease Health Care (Other)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO03-25-002
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2006-11

CONDITIONS: Prostate Cancer
Keywords: Hormone Refractory; Taxane Refractory
MeSH Terms: conditions — Prostatic Neoplasms | interventions — liposomal doxorubicin; Estramustine

INTERVENTIONS:
Drug: Doxil and Estramustine

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of the drug combination of Doxil (doxorubicin) and estramustine when used to treat prostate cancer that is resistant to hormones and to a chemotherapy type called taxanes.

The primary hypothesis is to reduce the measurable disease or prostate-specific antigen (PSA) level by at least 50% from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced, prostate cancer
* Patients must have evaluable disease that may be evaluated by PSA or measurement.
* Patients must be hormone refractory as defined in this protocol.
* Patients must be taxane refractory as defined in this protocol.
* Patients have had no prior chemotherapy other than a taxane or estramustine phosphate.
* Patients may have had prior radiation therapy (RT) if it has been >/= 4 weeks since completion.
* Patients on bisphosphonates may be included.
* Patients must be at least 18 years of age or older.
* Patients must have the ability to speak and understand English.
* Patients must have an ECOG performance status of 2 or less.
* Patients must have adequate bone marrow function: platelets > 100,000 cells/mm3; hemoglobin > 9.0 g/dL; and absolute neutrophil count (ANC) > 1,000 cells/mm3.
* Patients must have adequate renal function: creatinine < 2.5 mg/dL.
* Patients must have adequate liver function.
* Ejection fraction of > 50% within 42 days of first dose of study drug.
* Ability to complete the McGill-Melzack Pain Intensity Scale.

Exclusion Criteria:

* Patients with unstable medical conditions such as liver, renal dysfunctions, blood clots or heart disease.
* History of hypersensitivity to doxorubicin.
* History of class II cardiac disease or evidence of congestive heart failure.
* RT within the past 4 weeks of study entry or a radiopharmaceutical within the past 8 weeks of study entry.
* Prior malignancy within the past 5 years except for non-melanotic skin cancers.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-12

PRIMARY OUTCOMES:
Reduce the measurable disease and PSA level by at least 50%

SECONDARY OUTCOMES:
To determine safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Robert Drapkin, MD, Principal Investigator — Morton Plant Mease Health Care
Locations (1):
- Morton Plant Mease Health Care, Clearwater, Florida, United States